CLINICAL TRIAL: NCT03074305
Title: Randomized Controlled Trial for Comparison of Efficacy and Safety Between Drug-eluting Balloon and 2nd Generation Drug-Eluting Stent in Patients With In-Scaffold Restenosis of Bioresorbable Vascular Scaffold
Brief Title: DEB Versus 2nd Generation DES in Patients With In-Scaffold Restenosis of Bioresorbable Vascular Scaffold
Acronym: SMART-BRS-ISR
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: cannot use bioabsorbable scaffold
Sponsor: Samsung Medical Center (Other)
Responsible Party: Principal Investigator, Joo-Yong Hahn, Professor, Samsung Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BRS-ISR16453143
Record Dates: First submitted 2017-03-04; First posted 2017-03-08 (Actual); Last update posted 2024-04-22 (Actual); Status verified 2024-04

CONDITIONS: Coronary Artery Disease; Coronary Restenosis
Keywords: In-bioresorbable vascular scaffold restenosis; drug-eluting stent; drug-eluting balloon; bioresorbable scaffold
MeSH Terms: conditions — Coronary Artery Disease; Coronary Restenosis | interventions — Percutaneous Coronary Intervention

STUDY DESIGN:
Intervention Model Description: Prospective, open label, two-arm, randomized controlled trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- DEB strategy (Active Comparator): DEB procedure will be standardized in order to maximize drug delivery into target segment. Commercially available DEB will be used (Sequent Please, B Braun, Germany or Pantera Lux, Biotronik, German). The below requirements will be mandatorily recommended.
  1. Residual stenosis after lesion preparation : %DS <20%
  2. Delivery time : < 30 seconds
  3. Total inflation time : > at least 1 minute
  4. Previous BVS : DEB diameter ratio : > 1.0:1
  5. Maximum inflation pressure : at least above nominal pressure of DEB
  Interventions: Device: PCI for in-bioresorbable scaffold stenosis
- DES strategy (Active Comparator): The implantation of 2nd generation DES will be performed as universally recommended. In the DES group, the newest version of 2nd generation everolimus-eluting stent (Xience Alpine, Abbott Vascular, USA) will be recommended.
  Interventions: Device: PCI for in-bioresorbable scaffold stenosis

INTERVENTIONS:
Device: PCI for in-bioresorbable scaffold stenosis — In patients who have in-bioresorbable scaffold stenosis after bioresorbable scaffold implantation, PCI will performed according to the allocated arms
  1. DEB strategy
  2. DES strategy

SUMMARY:
The aim of the study is to compare angiographic outcomes following revascularization using drug-eluting balloon (DEB) versus 2nd generation drug-eluting stent (DES) in treatment of Bioresorbable Vascular Scaffold Restenosis.

DETAILED DESCRIPTION:
The bioresorbable vascular scaffold (BRS) has been emerged as new therapeutic option in percutaneous coronary intervention for coronary artery disease. Although 2nd generation drug-eluting stent (DES) has enhanced the efficacy and safety of DES, However, along with the widespread use of this newer generation DES in most clinical conditions, including high-risk patients with more complicated lesion profiles, ISR has continued to be a major concern, even in the era of newer generation DES. In this regards, the concept of BRS has introduced and has showed promising results. Nevertheless, previous reports showed that even BRS has not been free from restenosis, leading target lesion revascularization up to 7.4% during 3-year follow up. Currently, previous researches which comparedsafety and efficacy of treatment options for ISR lesion showed similar clinical outcomes following 2 representative options, namely, drug-eluting balloon or drug-eluting stent. In this regards, current European Society of Cardiology/European Association for Cardiothoracic Surgery (ESC/EACTS) guidelines recommend drug-eluting balloon (DEB) and 2nd generation DES as class IA recommendations for the treatment of BMS or DES-ISR. However, all the previous reports evaluated the ISR of metallic stents, and there has been no evidence for treatment option for BRS ISR.

Therefore, the Smart Angioplasty Research Team: Safety and Efficacy of Drug-Eluting Balloon versus 2nd Generation Drug-Eluting Stent in Treatment of In-Bioresorbable Vascular Scaffold Restenosis (SMART-BRS-ISR) trial will randomly allocate patients with BRS ISR into DEB or 2nd generation DES and compare safety and efficacy of both treatment options.

ELIGIBILITY:
Inclusion Criteria:

* Subject age 19-85 years old
* Patients with BRS ISR and presented with angina symptom or objective sign of inducible myocardial ischemia (one of the followings)

  1. Visual stenosis ≥50% in ISR segment with typical angina symptom (CCS class ≥II) or positive non-invasive stress tests
  2. ISR lesion with fractional flow reserve (FFR) ≤0.80
  3. Visual stenosis ≥70% in ISR segment (in the absence of above 2 components)
* Patients with BRS ISR which can be treated by DEB angioplasty or second generation DES implantation

Exclusion Criteria:

* Cardiogenic shock (Killip class IV) already at presentation or the completion of culprit PCI
* Intolerance to Aspirin, Clopidogrel, Plasugrel, Ticagrelor, Heparin, Bivaluridin, or Everolimus, Zotarolimus
* Patients with active bleeding or history of gastrointestinal or genitourinary major bleeding within 3-month
* Chronic kidney disease (serum creatinine ≥2.0mg/dL or estimated glomerular filtration rate <30ml/min)
* Known true anaphylaxis to contrast medium (not allergic reaction but anaphylactic shock)
* Non-cardiac co-morbid conditions are present with life expectancy <1 year or that may result in protocol non-compliance (per site investigator's medical judgment).
* In-segment edge restenosis without definite involvement of previous BRS edge
* Unwillingness or inability to comply with the procedures described in this protocol.

Ages: 19 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2017-03-08 (Actual); Primary Completion 2017-12-30 (Actual); Study Completion 2018-01-25 (Actual)

PRIMARY OUTCOMES:
Minimum lumen diameter (MLD) in BRS ISR lesion, post-PCI | 13-month after index procedure

SECONDARY OUTCOMES:
post-PCI FFR value | Immediate after index procedure
post-PCI MLD | Immediate after index procedure
minimum stent area (MSA) measured by intravascular ultrasound (IVUS) | Immediate after index procedure
minimum stent area measured by optical coherence tomography (OCT) | Immediate after index procedure
follow-up FFR | 13-month after index procedure
13-month follow-up minimal stent area measured by IVUS or OCT | 13-month after index procedure
  stratified analysis according to imaging modality
OCT findings in neoatherosclerotic tissue | 13-month after index procedure
  macrophage infiltration, presence of thin-cap fibrous neoatheroma (TCNA), patterns of neoatherosclerotic tissue (homogeneous, heterogeneous, layered, neoatherosclrotic), cap thickness
All-cause mortality | 12-month after index procedure
Cardiac death | 12-month after index procedure
Any myocardial infarction | 12-month after index procedure
12-month follow up any revascularization | 12-month after index procedure
Target vessel revascularization | 12-month after index procedure
Stent thrombosis | 12-month after index procedure
Major adverse cardiovascular events | 12-month after index procedure
  a composite of cardiac death, target-vessel MI, and target lesion revascularization

CONTACTS AND LOCATIONS:
Overall Officials: Joo-Yong Hahn, MD, PhD, Study Chair — Samsung Medical Center
Locations (1):
- Samsung Medical Center, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Yes
After publication of first manuscript and trial results, the de-identified data will be shared by permission of principle investigator, when asked